CLINICAL TRIAL: NCT05071118
Title: the Effect of Adding Pregabalin on the Onset and the Duration of Spinal Anesthesia and on the Postoperative Analgesia
Brief Title: The Efficacy of Pregabalin on the Duration of the Spinal Anesthesia and the Early Postoperative Pain After Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ismail Mohammed, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R71/2021
Record Dates: First submitted 2021-09-20; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregabalin group (Active Comparator): Two hours before surgery, the pregabalin patients (group P) received capsules containing 150mg of pregabalin in the ward then transferred to OR to receive spinal anesthesia before surgery.
  Interventions: Drug: Pregabalin 150mg
- placebo group (Active Comparator): The patients received placebo capsules in the ward Then transferred to OR to receive spinal anesthesia before surgery .
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin 150mg — pregabalin patients (group P) received capsules containing 150mg of pregabalin in the ward then transferred to OR to receive spinal anesthesia before surgery
  Arms: pregabalin group
Drug: Placebo — The patients received placebo capsules in the ward Then transferred to OR to receive spinal anesthesia before surgery .
  Arms: placebo group

SUMMARY:
the purpose of this study is to evaluate the effectiveness of administration of pregabalin 2 hours preoperatively on the onset and the duration of the spinal anesthesia in total knee arthroplasty and the role of pregabalin in postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* the ages of 40 and 70 years
* height 155-170 cm
* American Society of Anesthesiologists grade I or II .
* patients underwent total knee arthroplasty under spinal anesthesia

Exclusion Criteria:

* patients known to be allergic to any medicines.
* patients had a history of drug or alcohol abuse.
* patients were taking opioids or sedative medications,
* patients Inability to communicate with investigators to evaluate the postoperative pain
* patients were in need for postoperative ICU hospitalization .
* patients had a history of psychiatric conditions.
* Patients with a history of taking pregabalin or gabapentin .

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-03-21 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-08-25 (Actual)

PRIMARY OUTCOMES:
onset of spinal anaesthesia | three months
  seventy participants undergoing elective total knee arthroplasty under spinal anesthesia half of them took placebo and the other half took 150 mg pregabalin two hours before the procedure and calculate the time from the base line to the onset of anesthesia.
  Our primary outcome is to assess the onset of spinal anesthesia.
  to detect the onset of spinal anaesthesia

SECONDARY OUTCOMES:
recovery time | three months
  Recovery time from the sensory blockade (2-dermatome regression of anesthesia from the maximum level).
motor block duration | three months
  the time for return to Bromag 2 (the patient is able to move knees and ankles).
postoperative analgesia | three months.
  • Postoperative pain will be assessed by the patient using the visual analog scale in the first 24 hour(VAS, 0=no pain; 10=worst possible pain) every 2 hours up to 24 hours after the operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt